CLINICAL TRIAL: NCT06842602
Title: Evaluation of Gastric Volume and pH Changes in Gastroscopy Patients Using Chewing Gum and Candy: Prospective Randomized Double-Blind Study
Brief Title: Evaluation of Gastric Volume and pH Changes in Gastroscopy Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Mehmet Fatih Erol, m.d, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: 2023/07-11
Record Dates: First submitted 2025-02-19; First posted 2025-02-24 (Actual); Last update posted 2025-04-15 (Actual); Status verified 2025-04

CONDITIONS: Gastroscopy
Keywords: gastric pH; gastric residual volume; gastroscopy; candy; gum; preoperative fasting rules
MeSH Terms: interventions — Chewing Gum; Candy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group control (Active Comparator): strict fasting rules
  Interventions: Other: strict fasting rules
- Group gum (Active Comparator): chewed gum within 2 hours before the procedure
  Interventions: Other: gum
- Group candy (Active Comparator): consumed candy within 2 hours before the procedure
  Interventions: Other: candy

INTERVENTIONS:
Other: gum — chewed gum within 2 hours before the procedure
  Arms: Group gum
Other: candy — consumed candy within 2 hours before the procedure
  Arms: Group candy
Other: strict fasting rules — followed strict fasting rules
  Arms: Group control

SUMMARY:
Pulmonary aspiration is a rare but serious complication that can result in 57% mortality and 14% permanent damage. Fasting rules (solid foods 6-8 hours, clear liquids 2 hours) determined by anesthesia associations are applied to prevent pulmonary aspiration by reducing gastric volume. Gastric volume (≥ 0.5 mL/kg) and pH (<2.5) values are shown to be determinants in the occurrence of pulmonary complications .

DETAILED DESCRIPTION:
The hypothesis of this study was that preprocedure candy and chewing gum use may have no effects on gastric residual volume and pH. For this purpose, we analyzed the gastric residual volume and gastric pH values of patients who were given gum and candy before the procedure.

ELIGIBILITY:
Inclusion Criteria:

* ASA I-III,
* oriented
* cooperative
* scheduled for elective gastroscopy

Exclusion Criteria:

* body mass index is (BMI) >30 kg/m2,
* full stomach predicted patients (obstruction, stenosis, bleeding, ascites, urgency),
* patients with diabetes
* patients with who underwent bowel cleansing
* patients who did not want to give consent to participate

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
Gastric volume | baseline
  No washing was performed during the insertion and advancement of the endoscope. The entire gastric volume were aspirated into a scaled container (medbar collection container). The amount of collected samples was recorded .
Gastric pH measurements | baseline
  No washing was performed during the insertion and advancement of the endoscope. The entire gastric contents were aspirated into a scaled container (medbar collection container). The amount of collected samples was recorded and pH analysis (WTW inoLab® pH 7310 Table Type pH Meter) was performed.

SECONDARY OUTCOMES:
endoscopist satisfaction | baseline
  At the end of the procedure, endoscopist satisfaction (0=unsatisfied 1=abstained 2=satisfied) and procedure difficulty (0=easy 1=normal 2=difficult)
general procedure satisfaction | baseline
  Before discharge, general procedure satisfaction (0=unsatisfied, 1=abstained, 2=satisfied), product satisfaction (0=unsatisfied, 1=abstained, 2=satisfied), product effects (1=increase in hunger, 2=increase in thirst, 3=increase in dyspepsia, 4=abstained, 5= decrease in hunger, 6= decrease in thirst, 7= decrease in dyspepsia)
Complication | Perioperative

CONTACTS AND LOCATIONS:
Overall Officials: Mehmet fatih erol, M.D, Study Director — Bursa Yuksek ıhtısas tra; Füsun gözen, M.D, Study Director — Bursa Yuksek Ihtısas tranin and research hospital
Locations (1):
- Mehmet Fatih Erol, Bursa, Turkey (Türkiye)